CLINICAL TRIAL: NCT03801356
Title: Defining the Threshold Response of Lumbar Selective Nerve Root Block in Predicting Good Outcome Following Lumbar Foraminotomy
Brief Title: Threshold Response of Lumbar Selective Nerve Root Block in Predicting Good Outcome Following Lumbar Foraminotomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated early due to a number of concurrent issues: low enrollment, limited data and COVID-19.
Sponsor: The Cleveland Clinic (Other)
Collaborators: Lumbar Spine Research Society (Other)
Responsible Party: Principal Investigator, Michael Steinmetz, MD, Principal Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-718
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-06

CONDITIONS: Back Pain; Radiculopathy Lumbar; Degenerative Lumbar Spinal Stenosis
Keywords: back pain; lumbar spine pain; nerve root block; foraminotomy; radiculopathy; lumbar; foraminal stenosis
MeSH Terms: conditions — Back Pain; Low Back Pain; Radiculopathy

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled into a single treatment participant pool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Selective Nerve Root Block (Other): Patient will receive a Selective Nerve Root Block injection at the target level prior to surgical intervention.
  Interventions: Drug: Selective Nerve Root Block

INTERVENTIONS:
Drug: Selective Nerve Root Block — Prior to single level foraminotomy for lumbar foraminal stenosis, patients will undergo SNRB of the suspected nerve root. Patients will undergo surgery despite the response to injection. Patients will complete an ambulation assessment immediately before and after the injection. Distance and time will be noted. Patients will be called within 48 hours of injection to determine response to injection, and recorded as Pre-and Post-injection VAS leg as well as duration of the response. Patients will be seen at 6 weeks, 3,6, and 12 months post-surgery and outcome measured by VAS-leg, ODI, PDQ and EQ-5D scores. Data will be used to determine the ideal improvement in leg pain and duration of improvement, predicting a statistical and meaningful improvement in leg pain following foramintomy.

SUMMARY:
SNRB, as measured by the change in pain and objective functional ability, can solicit crucial information regarding a patient's clinical picture and can predict a patient's outcome post-surgery. By using the walk test as an objective functional assessment, the aim is to better standardize the threshold for a positive response to SNRB.

In summary, SNRB, despite utilized frequently in the diagnostic work-up with patients with lumbar radiculopathy, vary widely in their sensitivity and specificity. The reasons, as outlined above, are multifactorial. The proposed study aims to minimize the known limitations of these injections and prospectively define their positive and negative predictive value in a homogenous group of patients undergoing surgery for lumbar foraminal stenosis and radiculopathy. The design will define a threshold of response utilizing both subjective and objective measures and more accurately predict excellent results following surgery.

DETAILED DESCRIPTION:
The proposed study will identify the threshold response level that quantifies the predictive value of diagnostic SNRBs in patients who present with lumbar foraminal stenosis and radiculopathy. Specifically, the proposed study will address the question of whether there is a degree or length of response to SNRB, which predicts an excellent surgical outcome. The hypothesis is that diagnostic SNRBs, when performed correctly, are useful in localizing the level of involvement in LSS and improve the accuracy and efficacy of surgical intervention. Use of diagnostic SNRBs will thus be used to clarify the clinical picture, giving the surgeon the information to make the right decision to operate or not, and, in the case of operation, predicting the optimal level(s) for surgical intervention. In addition, the investigators plan to identify and fully characterize a standard threshold level and time of nerve block response that will optimize the accuracy, specificity, and sensitivity of SNRB in predicting surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-80
* Diagnosis of unilateral lower extremity radiculopathy due to degenerative foraminal stenosis
* Patients scheduled for an associated lumbar foraminotomy procedure
* Diagnosis of radiculopathy with imaging and/or clinical history or physical exam that does not demonstrate a clear neurogenic source of their pain
* Subjects must be available for the entire study duration (12 months)

Exclusion Criteria:

* Patients will be excluded if there is a clear correlation between imaging and radiculopathy
* Radiculopathy associated with trauma, tumor or infection. Non-radicular lower extremity pain will also be excluded
* Patients who cannot tolerate the SNRB without IV sedation
* Surgery requiring multi-level decompression and/or fusion
* Surgical indication for malignancy, injection or acute or emergency trauma
* History of major surgery within 3 months prior to enrollment
* Pregnant females
* Presence of severe acute, chronic medical or psychiatric condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Steinmetz, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Selective Nerve Root Block
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Selective Nerve Root Block
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Leg Pain Score
Description: Aim: 0-2 point improvement
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' (0) and 'pain as bad as it could be' (10). The patient is asked to mark their pain level on the line between the two endpoints. The distance and change between '0' and the mark then defines the subject's pain. This will be measured at each subject visit.
Time Frame: 12-months
Population: Paired T-Test was conducted to compare the change in VAS score from Baseline Visit to 12 Month Visit. Although 11 patients were consented and completed a Baseline Visit, only 7 patients had a 12 Month Visit. Analysis included the 7/11 patients that completed a 12 Month Visit that captured the VAS Leg Pain Score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Selective Nerve Root Block
Number analyzed (Participants) | 7
score on a scale | 1.14 (3.34)

2. Secondary Outcome: Oswestry Disability Index Questionnaire (ODI)
Description: Aim: 15-point improvement
  The Oswestry Disability Index (ODI) is one of the principal condition-specific outcome measures used in the management of spinal disorders. The ODI is the most commonly outcome measures in patients with low back pain.
  Structure / Content
  There are 10 questions. The questions are designed in a way that to realize how the back or leg pain is affecting the patient's ability to manage in everyday life.
  Scoring Method
  Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. The score can be multiplied by 2 to produce a percentage.
  If the FIRST statement is marked, the section score = 0, If the LAST statement is marked, it = 5
  Interpretation
  1.0%-20%: Minimal disability. Usually no treatment is indicated.
  2.20%-40% Moderate disability
  3.40%-60%: Severe disability
  4.60%-80%: Crippled
  5.80%-100%: These patients are either bed-bound or exaggerating their symptoms.
Time Frame: 12-Months
Population: Although 11 patients were consented and completed the Baseline Visit and 7/11 patients completed the VAS Leg Pain Score at 12 Month Visit, 0/11 patients completed an ODI Questionnaire at 12 Month Visit. Due to no patient completing the ODI at 12 Month Visit, no analysis was completed for this outcome measure.
Arm/Group | Selective Nerve Root Block
Number analyzed (Participants) | 0

3. Secondary Outcome: EQ-5D Questionnaire
Description: Aim: Improvement in quality of life
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The questionnaire also records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labeled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Time Frame: 12-Months
Population: Although 11 patients were consented and completed the Baseline Visit and 7/11 patients completed the VAS Leg Pain Score at 12 Month Visit, 0/11 patients completed an EQ-5D Questionnaire at 12 Month Visit. Due to no patient completing the EQ-5D at 12 Month Visit, no analysis was completed for this outcome measure.
Arm/Group | Selective Nerve Root Block
Number analyzed (Participants) | 0

4. Secondary Outcome: Pain Disability Questionnaire (PDQ)
Description: Aim: 26-point improvement
  The Pain Disability Questionnaire (PDQ) assesses perception of disability in relation to pain.
  PDQ scores: mild/moderate (0-70), severe (71-100), and extreme (101-150).
Time Frame: 12-months
Population: Although 11 patients were consented and completed the Baseline Visit and 7/11 patients completed the VAS Leg Pain Score at 12 Month Visit, 0/11 patients completed a PDQ Questionnaire at 12 Month Visit. Due to no patient completing the PDQ at 12 Month Visit, no analysis was completed for this outcome measure.
Arm/Group | Selective Nerve Root Block
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: For subjects who completed study, adverse events were collected during time on study, an average of 12 months. Adverse events were not collected after study termination.
Arm/Group | Selective Nerve Root Block
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
The study was terminated early due to a number of concurrent issues. We found it difficult to enroll patients. Many of the patients were from out of region and/or had presented with a concurrent spinal injection. A new study injection could not be ordered due to the aforementioned issues. We attempted to mitigate, but it proved to be difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT03801356/Prot_SAP_001.pdf